CLINICAL TRIAL: NCT01482143
Title: Sequential, Two-period Study to Assess the Pharmacokinetics, Safety & Tolerability of Single and Multiple Oral Doses of AFQ056 in Patients With FXS (Fragile X Syndrome) Aged 5-11 Years (Cohort 1) and 3-4 Years (Cohort 2)
Brief Title: Clinical Study to Assess the Pharmacokinetics, Safety and Tolerability of Single and Multiple Oral Doses of AFQ056 in Children With Fragile X Syndrome (FXS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAFQ056B2154; 2011-004867-65 (EudraCT Number)
Record Dates: First submitted 2011-11-21; First posted 2011-11-30 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2014-09

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; pharmacokinetics; safety and tolerability
MeSH Terms: conditions — Fragile X Syndrome | interventions — mavoglurant

ARMS (1):
- All Study subjects (Experimental)
  Interventions: Drug: AFQ056

INTERVENTIONS:
Drug: AFQ056

SUMMARY:
The aim of this study is to characterize the pharmacokinetics and safety/tolerability of AFQ056 in children with Fragile X Syndrome(FXS)

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of FXS
* At Screening and first baseline, vital signs, body weight and body mass index (BMI) must be age-specific within normal ranges.

Exclusion Criteria:

* Use of any other investigational drug within 30 days or 5 half-lives (whichever is longer) of the investigational drug prior to screening until end of study visit.
* History of hypersensitivity to AFQ056 or any mGluR antagonist.
* Female patients who are confirmed or suspected to be sexually active.
* History or presence of any clinically significant disease of any major system organ class, within the past 2 years prior to screening including but not limited to psychiatric, neurological, cardiovascular, endocrine, metabolic, renal, or gastrointestinal disorders (except for typical features of FXS).
* Smokers.
* Loss of ≥10% of total blood volume within 8 weeks (or less if required for this age group and/or by local regulation) prior to dosing or longer if required for this age group and/or by local regulation.
* Significant illness that did not completely resolve at least four weeks prior to the first baseline visit.
* Any abnormal laboratory values at screening or first baseline that are in the opinion of the investigator clinically significant and may jeopardize the safety of the study subject.
* Use of (or use within at least 5 half lives before dosing) concomitant medications that are strong/moderate inhibitors or inducers of CYP1A1/2, CYP2C9/19 or CYP3A4
* History or presence of Hepatitis B/C or HIV at screening

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The area under the plasma (or serum or blood) concentration-time curve from time zero to infinity [mass x time / volume] (AUCinf) | Time Frame: Day 1 (period 1): 0.5, 2, 4, 8, 12, 24 hours post-dose; Day 7 (period 2): pre-dose; 0.5, 2, 4, 8 hours post dose
The area under the plasma (or serum or blood) concentration-time curve from time zero to the time of the last quantifiable concentration [mass x time / volume] (AUClast) | Time Frame: Day 1 (period 1): 0.5, 2, 4, 8, 12, 24 hours post-dose; Day 7 (period 2): pre-dose; 0.5, 2, 4, 8 hours post dose
Maximum observed plasma concentration (Cmax) | Time Frame: Day 1 (period 1): 0.5, 2, 4, 8, 12, 24 hours post-dose; Day 7 (period 2): pre-dose; 0.5, 2, 4, 8 hours post dose

SECONDARY OUTCOMES:
Physical examination | Screening: once anytime between Day -30 and Day -1; once anytime between 24-72 hours after Day 7
Vital signs and body measurements | Screening: once anytime between Day -30 and Day -1; once anytime between 24-72 hours after Day 7
Electrocardiograms | Screening: once anytime between Day -30 and Day -1; once anytime between 24-72 hours after Day 7
hematology | Screening: once anytime between Day -30 and Day -1; once anytime between 24-72 hours after Day 7
blood chemistry | Screening: once anytime between Day -30 and Day -1; once anytime between 24-72 hours after Day 7
neurological examination | Screening: once anytime between Day -30 and Day -1; once on Day 7
Adverse events (AE) monitoring | During the study (total of approximately 32 days) and 3 days after study completion
Serious adverse events (SAE) monitoring | During the study (total of approximately 32 days) and 30 days after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (3):
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Nashville, Tennessee
- Novartis Investigative Site, Sant Cugat del Vallès, Catalonia, Spain

REFERENCES:
- See also: Results for CAFQ056B2154 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=11925